CLINICAL TRIAL: NCT01656408
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8150
Brief Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8150 (MK-8150-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8150-002; 2012-002596-34 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-08-03 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Isolated Systolic Hypertension
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension | interventions — MK-8150

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Panel A: Mild/Moderate Hypertension (Experimental): MK-8150 or matching placebo once daily, capsules, oral, for 10 days
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel B: Mild/Moderate Hypertension (Experimental): MK-8150 or matching placebo once daily, capsules, oral, for 10 days
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel C: Mild/Moderate Hypertension (Experimental): MK-8150 or matching placebo once daily, capsules, oral, for 10 days
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel D: Mild/Moderate Hypertension (Experimental): MK-8150 or matching placebo once daily, capsules, oral, for 10 days
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel E-Elderly (Experimental): Single dose of MK-8150 or placebo on Study Day 1 followed by a wash-out of at least 5 days, then MK-8150 or placebo once daily at a lower dose for 10 days
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel F - Elderly (Experimental): Single dose of MK-8150 or placebo on Study Day 1 followed by a wash-out of at least 5 days, then MK-8150 or placebo once daily at a lower dose for 10 days
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel G - Healthy - Dose Titration (Experimental): MK-8150 or matching placebo will be administered once daily for 28 days. Dose may be adjusted on Day 8, Day 15, and Day 22.
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel H - Crossover (Experimental): MK-8150 or matching placebo for 10 consecutive days in 2-period crossover with minimum 3 weeks washout period between the 2 treatment periods
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel I - Dose Titration (Experimental): MK-8150 or matching placebo will be administered once daily for 28 days. Dose may be adjusted on Day 8, Day 15, and Day 22.
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150
- Panel J - Dose Titration (Experimental): MK-8150 or matching placebo will be administered once daily for 28 days. Dose may be adjusted on Day 8, Day 15, and Day 22.
  Interventions: Drug: MK-8150; Drug: Placebo for MK-8150

INTERVENTIONS:
Drug: MK-8150
Drug: Placebo for MK-8150

SUMMARY:
This randomized, double-blind, placebo-controlled, multiple-rising-dose study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of MK-8150 in healthy young men, in male participants with mild to moderate hypertension, in elderly male and female participants with mild to moderate hypertension, and in male and female participants with resistant hypertension. A primary study hypothesis is that there is at least one dose that does not increase heart rate (HR) to a clinically meaningful extent in male participants with mild to moderate hypertension and in elderly participants with mild to moderate hypertension on either Day 1 or the last Day of multiple dosing (Daylast), as measured by Time-weighted Average Across 24 hours (TWA0-24hrs). The hypothesis is met if mean increase (MK-8150 - placebo) in TWA0-24hrs HR in the identified groups is ≤15 beats per minute on Day 1 and Daylast.

DETAILED DESCRIPTION:
Ten panels (Panels A-J), consisting of 103 participants in total, will be randomized to receive either MK-8150 or matching placebo.

Males (18 to 55 years of age, inclusive) with mild to moderate hypertension will be randomized in Panels A-D and will receive either MK-8150 or placebo as once daily treatment for 10 consecutive days.

Elderly males and females (65 to 80 years of age, inclusive) with mild to moderate hypertension will be included in Panels E and F and will receive a single dose of either MK-8150 or placebo on Study Day 1 followed by at least 5 days of wash-out before proceeding to once daily treatment of the same randomized treatment at a lower dose for 10 consecutive days.

Participants 18 to 65 years of age with resistant hypertension will be enrolled in Panels H and will receive in randomized sequences of MK-8150/placebo or placebo/MK-8150 in 2 treatment periods. There will be a minimum 3 weeks washout period between the 2 treatment periods in Panel H.

Healthy males (18 to 55 years of age, inclusive) will be enrolled in Panel G and will receive MK-8150 or matching placebo once daily for 28 days. Participants randomized to MK-8150 in Panel G who meet all of the dose-escalation criteria and have not met any of the hemodynamic stopping criteria will be eligible for dose increases on Day 8, Day 15, and Day 22. If dose escalation criteria are not met (or if the Investigator or Sponsor elects not to increase the dose), then the participant will continue on the current dose and will be eligible for a dose increase at the next dose-escalation decision day if all dose-escalation criteria are met at that time.

Male participants (18 to 65 years of age, inclusive) with mild to moderate hypertension will be randomized in Panels I and J. In each panel, 18 participants will receive either MK-8150 or matching placebo as once daily treatment for up to 28 consecutive days. Participants who are randomized to placebo will receive placebo throughout the study. On Days 8, 15 and 22 in both Panels I and J, participants will be eligible for dose-escalation, down-dosing, or continuing their current dose depending on their hemodynamic status. Participants in Panels I and J who meet down-dosing criteria at any time during the study will have their doses reduced to the previous well-tolerated dose level until the next dose-escalation decision day, or through the end of the study, whichever is first.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive male participant between 18 to 55 years of age for Panels A to D; hypertensive male or female of non-childbearing potential between 65 to 80 years of age for Panels E and F; healthy males between 18 to 55 years of age for Panel G; hypertensive male or non-childbearing potential female between 18 to 65 years of age (inclusive) for Panel H; hypertensive male between 18 to 65 years of age for Panels I and J
* Body Mass Index (BMI) ≤ 33 kg/m^2
* In good age appropriate health
* No history of clinically significant cardiac disease
* Nonsmoker and/or has not used nicotine or nicotine-containing products for at least 6 months

Exclusion Criteria:

* Mentally or legally incapacitated, has significant emotional problems or has a history of a clinically significant psychiatric disorder over the last 5 years
* History of stroke, chronic seizures, or a relevant major neurological disorder
* History of neoplastic disease (cancer)
* Unable to refrain from or anticipates the use of any medication, including any non-steroidal anti-inflammatory drug (NSAID) and aspirin-containing products, prescription and non-prescription drugs or herbal remedies for 2 weeks prior to study start up to end of study
* Anticipates using erectile dysfunction medications during the study
* Uses or anticipates using organic nitrates during the course of the study (e.g. nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, pentaerythritol)
* Consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Has had major surgery, donated or lost 1 unit of blood or participated in another investigational study within 4 weeks
* History of significant multiple and/or severe allergies (including latex allergy)
* Current regular user (including recreational use) of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-05-03 (Actual); Study Completion 2013-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Knox CD, de Kam PJ, Azer K, Wong P, Ederveen AG, Shevell D, Morabito C, Meehan AG, Liu W, Reynders T, Denef JF, Mitselos A, Jonathan D, Gutstein DE, Mitra K, Sun SY, Lo MM, Cully D, Ali A. Discovery and Clinical Evaluation of MK-8150, A Novel Nitric Oxide Donor With a Unique Mechanism of Nitric Oxide Release. J Am Heart Assoc. 2016 Aug 25;5(9):e003493. doi: 10.1161/JAHA.116.003493. PMID 27561272
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=8150-002&kw=8150-002&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel A - Participants With Mild to Moderate Hypertension: 6 participants were randomly assigned to receive MK-8150 5 mg once daily and 2 participants were randomly assigned to receive placebo once daily for 10 days
- Panel B - Participants With Mild to Moderate Hypertension: 6 participants were randomly assigned to receive MK-8150 10 mg once daily and 2 participants were randomly assigned to receive placebo once daily for 10 days
- Panel C - Participants With Mild to Moderate Hypertension: 6 participants were randomly assigned to receive MK-8150 20 mg once daily and 2 participants were randomly assigned to receive placebo once daily for 10 days
- Panel D - Participants With Mild to Moderate Hypertension: 5 participants were randomly assigned to receive MK-8150 15 mg once daily and 2 participants were randomly assigned to receive placebo once daily for 10 days
- Panel E - Elderly Participants With Mild/Moderate Hypertension: 6 participants were randomly assigned to receive a single dose of MK-8150 3 mg on Day 1 and to also receive MK-8150 2 mg once daily on Days 6-15 (10 days of multiple dose administration); 3 participants were randomly assigned to receive placebo (single dose) on Day 1 and once daily on Days 6-15
- Panel F - Elderly Participants With Mild/Moderate Hypertension: 6 participants were randomly assigned to receive a single dose of MK-8150 6 mg on Day 1 and to also receive MK-8150 4 mg once daily on Days 6-15 (10 days of multiple dose administration); 3 participants were randomly assigned to receive placebo (single dose) on Day 1 and once daily on Days 6-15
- Panel G - Healthy Participants: 8 participants were randomly assigned to receive MK-8150 once daily as follows: 20 mg (Days 1-7), 30 mg (Days 8-14), 40 mg (Days 15-21), 60 mg (Days 22-28); 2 participants were randomly assigned to receive placebo once daily on Days 1-28. Dose administered could be increased or decreased based on defined criteria
- Panel H - Participants With Resistant Hypertension: In Panel with crossover design, 4 participants were randomly assigned to receive active drug (MK-8150) in Period 1 and placebo in Period 2 and 4 participants were randomly assigned to receive placebo in Period 1 and active drug in Period 2. Active drug regimen was MK-8150 once daily as follows: 10 mg (Days 1-2), 20 mg (Days 3-10); placebo regimen was placebo once daily on Days 1-10
- Panel I - Participants With Mild to Moderate Hypertension: 12 participants were randomly assigned to receive MK-8150 once daily as follows: 5 mg (Days 1-7), 10 mg (Days 8-14), 20 mg (Days 15-21), 40 mg (Days 22-28); 6 participants were randomly assigned to receive placebo once daily on Days 1-28. Dose administered could be increased or decreased based on defined criteria
- Panel J - Participants With Mild to Moderate Hypertension: 12 participants were randomly assigned to receive MK-8150 once daily as follows: 10 mg (Days 1-7), 20 mg (Days 8-28); 6 participants were randomly assigned to receive placebo once daily on Days 1-28. Dose administered could be increased or decreased based on defined criteria
Period: Overall Study
Arm/Group | Panel A - Participants With Mild to Moderate Hypertension | Panel B - Participants With Mild to Moderate Hypertension | Panel C - Participants With Mild to Moderate Hypertension | Panel D - Participants With Mild to Moderate Hypertension | Panel E - Elderly Participants With Mild/Moderate Hypertension | Panel F - Elderly Participants With Mild/Moderate Hypertension | Panel G - Healthy Participants | Panel H - Participants With Resistant Hypertension | Panel I - Participants With Mild to Moderate Hypertension | Panel J - Participants With Mild to Moderate Hypertension
Started | 8 | 8 | 8 | 7 | 9 | 9 | 10 | 8 | 18 | 18
Completed | 7 | 8 | 6 | 7 | 8 | 7 | 9 | 7 | 16 | 15
Not Completed | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A - Participants With Mild to Moderate Hypertension | Panel B - Participants With Mild to Moderate Hypertension | Panel C - Participants With Mild to Moderate Hypertension | Panel D - Participants With Mild to Moderate Hypertension | Panel E - Elderly Participants With Mild/Moderate Hypertension | Panel F - Elderly Participants With Mild/Moderate Hypertension | Panel G - Healthy Participants | Panel H - Participants With Resistant Hypertension | Panel I - Participants With Mild to Moderate Hypertension | Panel J - Participants With Mild to Moderate Hypertension | Total
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 9 | 9 | 10 | 8 | 18 | 18 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (6.3) | 41.3 (10.8) | 42.0 (11.4) | 42.7 (10.8) | 72.6 (4.2) | 69.9 (2.5) | 41.5 (11.2) | 58.1 (5.6) | 51.5 (8.5) | 54.8 (9.6) | 52.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 4 | 5 | 0 | 3 | 0 | 0 | 12
  Male | 8 | 8 | 8 | 7 | 5 | 4 | 10 | 5 | 18 | 18 | 91
Central Systolic Blood Pressure (cSBP) [Mean (Standard Deviation); unit: mm Hg] — N for Panel H = 7; N for Total = 102
  mm Hg | 141 (15) | 126 (10) | 127 (16) | 126 (7) | 143 (11) | 144 (11) | 103 (11) | 130 (12) | 133 (10) | 136 (12) | 131 (16)
Heart Rate (HR) [Mean (Standard Deviation); unit: beats per minute] — N for Panel H = 7; N for Total = 102
  beats per minute | 65 (14) | 63 (7) | 66 (12) | 61 (10) | 59 (11) | 68 (9) | 54 (7) | 63 (9) | 62 (10) | 66 (9) | 63 (10)
Augmentation Index (AIx) [Mean (Standard Deviation); unit: percent] — N for Panel H = 7; N for Total = 102
  percent | 23 (8) | 13 (12) | 11 (18) | 10 (12) | 31 (7) | 30 (6) | 5 (15) | 20 (11) | 19 (9) | 23 (7) | 19 (13)
Central Diastolic Blood Pressure (cDBP) [Mean (Standard Deviation); unit: mm Hg] — N for Panel H = 7; N for Total = 102
  mm Hg | 93 (5) | 87 (8) | 87 (10) | 87 (7) | 84 (7) | 86 (11) | 73 (9) | 85 (8) | 89 (6) | 90 (11) | 87 (10)
Peripheral Systolic Blood Pressure (pSBP) [Mean (Standard Deviation); unit: mm Hg] — N for Panel H = 7; N for Total = 102
  mm Hg | 150 (12) | 137 (7) | 142 (17) | 139 (5) | 147 (10) | 151 (9) | 117 (7) | 141 (11) | 145 (9) | 147 (10) | 142 (13)
Peripheral Diastolic Blood Pressure (pDBP) [Mean (Standard Deviation); unit: mm Hg] — N for Panel H = 7; N for Total = 102
  mm Hg | 92 (6) | 86 (9) | 90 (10) | 86 (7) | 82 (5) | 86 (11) | 72 (9) | 84 (8) | 89 (6) | 90 (10) | 86 (10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study drug, is also an AE. The 8 crossover Panel H participants are represented in both Panel H - MK-8150 10/20 mg column and Placebo (Panel A - J) column.
Time Frame: Up to 14 days after the last dose (Up to approximately 42 days, excluding pre-dose/screening period)
Population: All participants who received at least one dose of study drug
Measure: Number; unit: participants
Groups:
- Panel A - MK-8150 5 mg: MK-8150 5 mg once daily for 10 days
- Panel B - MK-8150 10 mg: MK-8150 10 mg once daily for 10 days
- Panel C - MK-8150 20 mg: MK-8150 20 mg once daily for 10 days
- Panel D - MK-8150 15 mg: MK-8150 15 mg once daily for 10 days
- Panel E - MK-8150 3/2 mg: Single dose of MK-8150 3 mg on Day 1 and MK-8150 2 mg once daily on Days 6-15
- Panel F - MK-8150 6/4 mg: Single dose of MK-8150 6 mg on Day 1 and MK-8150 4 mg once daily on Days 6-15
- Panel G - MK-8150 20/30/40/60 mg: MK-8150 once daily as follows: 20 mg (Days 1-7), 30 mg (Days 8-14), 40 mg (Days 15-21), 60 mg (Days 22-28)
- Panel H - MK-8150 10/20 mg: MK-8150 once daily as follows: 10 mg (Days 1-2), 20 mg (Days 3-10)
- Panel I - MK-8150 5/10/20/40 mg: MK-8150 once daily as follows: 5 mg (Days 1-7), 10 mg (Days 8-14), 20 mg (Days 15-21), 40 mg (Days 22-28)
- Panel J - MK-8150 10/20 mg: MK-8150 once daily as follows: 10 mg (Days 1-7), 20 mg (Days 8-28)
- Placebo (Panel A - J): Combines participants who received placebo in all panels
- Post Study: All enrolled participants, presents AEs with onset after safety follow-up period after last dose of study drug
- Screening: All enrolled participants, presents AEs with onset before first dose of study drug
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel E - MK-8150 3/2 mg | Panel F - MK-8150 6/4 mg | Panel G - MK-8150 20/30/40/60 mg | Panel H - MK-8150 10/20 mg | Panel I - MK-8150 5/10/20/40 mg | Panel J - MK-8150 10/20 mg | Placebo (Panel A - J) | Post Study | Screening
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 8 | 8 | 12 | 12 | 36 | 103 | 103
participants | 4 | 5 | 6 | 3 | 4 | 3 | 7 | 6 | 12 | 10 | 24 | 1 | 12

2. Primary Outcome: Number of Participants Discontinued From Study Drug Due to Meeting Hemodynamic Stopping Rules
Description: Hemodynamic criteria for stopping drug dosing were applied (any of the following, obtained resting and if present for ≥1 hour, unless noted). For all Panels: HR >120 bpm; SBP ≥180 mm Hg (Panels A-D/G-J) and ≥175 mm Hg (Panels E-F); DBP ≥110 mm Hg; DBP <50 mm Hg; SBP <90 mm Hg or participant placed in Trendelenburg position. For Panels A-H: HR increase over identified baseline of ≥25 beats per minute; SBP reduction >30 mm Hg versus identified baseline; >20 mm Hg drop in SBP and >20 beats per minute rise in HR observed together versus identified baselines; >30 mm Hg drop in orthostatic SBP and >30 beats per minute rise in orthostatic HR observed together. For Panels I-J, any of the following-down dosing criteria if still present 24 hours after dose decrease: HR increase ≥20 beats per minute versus identified baseline; SBP reduction >30 mm Hg versus identified baseline; SBP <100 mm Hg; >30 mm Hg drop in orthostatic SBP and >30 beats per minute rise in orthostatic HR observed together.
Time Frame: Up to 28 days
Population: All participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel E - MK-8150 3/2 mg | Panel F - MK-8150 6/4 mg | Panel G - MK-8150 20/30/40/60 mg | Panel H - MK-8150 10/20 mg | Panel I - MK-8150 5/10/20/40 mg | Panel J - MK-8150 10/20 mg | Placebo (Panel A - J)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 8 | 8 | 12 | 12 | 36
participants | 3 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 3 | 0

3. Primary Outcome: Change From Baseline in Time-weighted Average Across 24 Hours (TWA0-24hrs) cSBP in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel A/B/C/D)
Description: cSBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cSBP value by that cSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel A/B/C/D - Placebo: Placebo once daily for 10 days, combining participants who received placebo in Panels A, B, C and D
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel A/B/C/D - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8
mm Hg
  Day 1 (N = 6, 6, 6, 5, 8) | -5.3 (2.6) | -15.3 (2.4) | -19.5 (2.4) | -12.8 (2.3) | -5.4 (2.3)
  Day 10 (N = 5, 6, 4, 5, 8) | -6.2 (3.4) | -13.9 (1.0) | -18.4 (1.9) | -12.1 (3.7) | -9.7 (3.0)
Statistical Analysis 1: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.978, Mixed Models Analysis; Least Squares (LS) Mean Difference = 0.1, 90% CI 2-sided [-6.4 to 6.6], Standard Error of Mean 3.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; LS Mean Difference = -9.9, 90% CI 2-sided [-15.4 to -4.5], Standard Error of Mean 3.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.000, Mixed Models Analysis; LS Mean Difference = -14.1, 90% CI 2-sided [-19.8 to -8.4], Standard Error of Mean 3.3 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; LS Mean Difference = -7.4, 90% CI 2-sided [-13.0 to -1.9], Standard Error of Mean 3.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.484, Mixed Models Analysis; LS Mean Difference = 3.5, 90% CI 2-sided [-4.9 to 11.9], Standard Error of Mean 4.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 6: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.169, Mixed Models Analysis; LS Mean Difference = -4.2, 90% CI 2-sided [-9.3 to 0.9], Standard Error of Mean 3.0 — Difference is MK-8150 dose - placebo
Statistical Analysis 7: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; LS Mean Difference = -8.7, 90% CI 2-sided [-14.9 to -2.6], Standard Error of Mean 3.6 — Difference is MK-8150 dose - placebo
Statistical Analysis 8: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.605, Mixed Models Analysis; LS Mean Difference = -2.4, 90% CI 2-sided [-10.4 to 5.5], Standard Error of Mean 4.6 — Difference is MK-8150 dose - placebo

4. Primary Outcome: Change From Baseline in TWA0-24hrs HR in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel A/B/C/D)
Description: HR was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all HR values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each HR value by that HR value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified HR value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel A/B/C/D - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8
beats per minute
  Day 1 (N = 6, 6, 6, 5, 8) | 0.0 (3.7) | -7.2 (2.5) | -12.3 (2.4) | -4.0 (3.2) | -1.9 (1.3)
  Day 10 (N = 5, 6, 4, 5, 8) | -3.6 (1.3) | -5.5 (2.0) | -10.5 (1.6) | -1.0 (2.4) | -2.1 (2.0)
Statistical Analysis 1: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.635, Mixed Models Analysis; LS Mean Difference = 1.9, 90% CI 2-sided [-4.9 to 8.7], Standard Error of Mean 3.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.077, Mixed Models Analysis; LS Mean Difference = -5.3, 90% CI 2-sided [-10.1 to -0.4], Standard Error of Mean 2.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference = -10.4, 90% CI 2-sided [-15.0 to -5.7], Standard Error of Mean 2.7 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.556, Mixed Models Analysis; LS Mean Difference = -2.1, 90% CI 2-sided [-8.0 to 3.9], Standard Error of Mean 3.5 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.527, Mixed Models Analysis; LS Mean Difference = -1.5, 90% CI 2-sided [-5.5 to 2.5], Standard Error of Mean 2.3 — Difference is MK-8150 dose - placebo
Statistical Analysis 6: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.234, Mixed Models Analysis; LS Mean Difference = -3.4, 90% CI 2-sided [-8.1 to 1.4], Standard Error of Mean 2.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 7: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; LS Mean Difference = -8.4, 90% CI 2-sided [-12.7 to -4.1], Standard Error of Mean 2.5 — Difference is MK-8150 dose - placebo
Statistical Analysis 8: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.726, Mixed Models Analysis; LS Mean Difference = 1.1, 90% CI 2-sided [-4.2 to 6.5], Standard Error of Mean 3.1 — Difference is MK-8150 dose - placebo

5. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel E)
Description: cSBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cSBP value by that cSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline for Day 1 was Day 1 pre-dose value; Baseline for Day 6-15 was Day 6 pre-dose value.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel E - Placebo: Placebo (single dose) on Day 1 and once daily on Days 6-15
Arm/Group | Panel E - MK-8150 3/2 mg | Panel E - Placebo
Number analyzed (Participants) | 6 | 3
mm Hg
  Day 1 (N = 6, 3) | -16.3 (3.3) | -15.5 (3.2)
  Day 6 (N = 5, 3) | -11.8 (3.6) | -15.5 (7.3)
  Day 15 (N = 5, 3) | -10.6 (3.9) | -16.9 (5.9)
Statistical Analysis 1: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 1; Test type: Superiority or Other; p = 0.855, Mixed Models Analysis; LS Mean Difference = -0.9, 90% CI 2-sided [-9.0 to 7.3], Standard Error of Mean 4.5 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 6; Test type: Superiority or Other; p = 0.658, Mixed Models Analysis; LS Mean Difference = 3.7, 90% CI 2-sided [-10.8 to 18.1], Standard Error of Mean 8.1 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 15; Test type: Superiority or Other; p = 0.392, Mixed Models Analysis; LS Mean Difference = 6.3, 90% CI 2-sided [-6.3 to 18.9], Standard Error of Mean 7.1 — Difference is MK-8150 dose - placebo

6. Primary Outcome: Change From Baseline in TWA0-24hrs HR in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel E)
Description: HR was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all HR values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each HR value by that HR value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified HR value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline for Day 1 was Day 1 pre-dose value; Baseline for Day 6-15 was Day 6 pre-dose value.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel E - MK-8150 3/2 mg | Panel E - Placebo
Number analyzed (Participants) | 6 | 3
beats per minute
  Day 1 (N = 6, 3) | 0.5 (1.2) | 2.0 (2.2)
  Day 6 (N = 5, 3) | 1.6 (0.8) | 0.8 (0.3)
  Day 15 (N = 5, 3) | 2.5 (1.3) | 0.7 (1.3)
Statistical Analysis 1: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 1; Test type: Superiority or Other; p = 0.563, Mixed Models Analysis; LS Mean Difference = -1.5, 90% CI 2-sided [-6.0 to 3.0], Standard Error of Mean 2.5 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 6; Test type: Superiority or Other; p = 0.381, Mixed Models Analysis; LS Mean Difference = 0.8, 90% CI 2-sided [-0.8 to 2.5], Standard Error of Mean 0.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 15; Test type: Superiority or Other; p = 0.387, Mixed Models Analysis; LS Mean Difference = 1.8, 90% CI 2-sided [-1.7 to 5.2], Standard Error of Mean 2.0 — Difference is MK-8150 dose - placebo

7. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel F)
Description: as for outcome 5
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel F - Placebo: Placebo (single dose) on Day 1 and once daily on Days 6-15
Arm/Group | Panel F - MK-8150 6/4 mg | Panel F - Placebo
Number analyzed (Participants) | 6 | 3
mm Hg
  Day 1 (N = 6, 3) | -16.1 (3.6) | -20.5 (3.1)
  Day 6 (N = 6, 3) | -17.2 (3.9) | -24.6 (2.7)
  Day 15 (N = 4, 3) | -20.8 (3.6) | -23.8 (3.6)
Statistical Analysis 1: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 1; Test type: Superiority or Other; p = 0.357, Mixed Models Analysis; LS Mean Difference = 4.5, 90% CI 2-sided [-3.9 to 12.8], Standard Error of Mean 4.7 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 6; Test type: Superiority or Other; p = 0.150, Mixed Models Analysis; LS Mean Difference = 7.4, 90% CI 2-sided [-1.2 to 15.9], Standard Error of Mean 4.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 15; Test type: Superiority or Other; p = 0.578, Mixed Models Analysis; LS Mean Difference = 3.0, 90% CI 2-sided [-6.3 to 12.3], Standard Error of Mean 5.2 — Difference is MK-8150 dose - placebo

8. Primary Outcome: Change From Baseline in TWA0-24hrs HR in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel F)
Description: as for outcome 6
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel F - MK-8150 6/4 mg | Panel F - Placebo
Number analyzed (Participants) | 6 | 3
beats per minute
  Day 1 (N = 6, 3) | -1.2 (1.7) | -1.5 (2.4)
  Day 6 (N = 6, 3) | -0.2 (1.7) | -2.1 (3.3)
  Day 15 (N = 4, 3) | -1.6 (1.5) | -5.8 (1.1)
Statistical Analysis 1: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 1; Test type: Superiority or Other; p = 0.942, Mixed Models Analysis; LS Mean Difference = 0.2, 90% CI 2-sided [-5.1 to 5.5], Standard Error of Mean 3.0 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 6; Test type: Superiority or Other; p = 0.627, Mixed Models Analysis; LS Mean Difference = 1.9, 90% CI 2-sided [-4.8 to 8.5], Standard Error of Mean 3.7 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 15; Test type: Superiority or Other; p = 0.046, Mixed Models Analysis; LS Mean Difference = 4.3, 90% CI 2-sided [0.9 to 7.6], Standard Error of Mean 1.9 — Difference is MK-8150 dose - placebo

9. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Healthy Male Participants Administered Multiple Doses of MK-8150 and Placebo (Panel G)
Description: as for outcome 3
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel G - Placebo: Placebo once daily on Days 1-28
Arm/Group | Panel G - MK-8150 20/30/40/60 mg | Panel G - Placebo
Number analyzed (Participants) | 8 | 2
mm Hg
  Day 1 (N = 8, 2) | -8.0 (1.7) | 2.8 (3.3)
  Day 28 (N = 7, 2) | -8.3 (2.2) | -2.3 (1.0)
Statistical Analysis 1: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 1; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; LS Mean Difference = -10.8, 90% CI 2-sided [-18.0 to -3.6], Standard Error of Mean 3.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 28; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis; LS Mean Difference = -6.0, 90% CI 2-sided [-11.0 to -1.1], Standard Error of Mean 2.6 — Difference is MK-8150 dose - placebo

10. Primary Outcome: Change From Baseline in TWA0-24hrs HR in Healthy Male Participants Administered Multiple Doses of MK-8150 and Placebo (Panel G)
Description: as for outcome 4
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel G - MK-8150 20/30/40/60 mg | Panel G - Placebo
Number analyzed (Participants) | 8 | 2
beats per minute
  Day 1 (N = 8, 2) | -1.1 (1.4) | -1.1 (1.4)
  Day 8 (N = 8, 2) | 0.5 (2.1) | 0.8 (1.4)
  Day 15 (N = 7, 2) | 2.3 (2.4) | 0.2 (1.4)
  Day 22 (N = 7, 2) | 0.8 (1.6) | 1.1 (1.6)
  Day 28 (N = 7, 2) | 1.8 (2.0) | 0.5 (1.4)
Statistical Analysis 1: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 1; Test type: Superiority or Other; p = 0.999, Mixed Models Analysis; LS Mean Difference = 0.0, 90% CI 2-sided [-4.4 to 4.4], Standard Error of Mean 2.6 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 8; Test type: Superiority or Other; p = 0.934, Mixed Models Analysis; LS Mean Difference = -0.3, 90% CI 2-sided [-5.7 to 5.2], Standard Error of Mean 3.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 15; Test type: Superiority or Other; p = 0.547, Mixed Models Analysis; LS Mean Difference = 2.1, 90% CI 2-sided [-3.7 to 7.9], Standard Error of Mean 3.4 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 22; Test type: Superiority or Other; p = 0.906, Mixed Models Analysis; LS Mean Difference = -0.3, 90% CI 2-sided [-5.2 to 4.5], Standard Error of Mean 2.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 28; Test type: Superiority or Other; p = 0.682, Mixed Models Analysis; LS Mean Difference = 1.3, 90% CI 2-sided [-4.0 to 6.6], Standard Error of Mean 3.1 — Difference is MK-8150 dose - placebo

11. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel H)
Description: cSBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cSBP value by that cSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value (determined separately in each period).
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel H - Placebo: Placebo once daily on Days 1-10
Arm/Group | Panel H - MK-8150 10/20 mg | Panel H - Placebo
Number analyzed (Participants) | 7 | 8
mm Hg
  Day 1 (N = 7, 8) | -10.1 (1.8) | -4.5 (1.8)
  Day 10 (N = 6, 8) | -7.7 (2.2) | -1.8 (1.0)
Statistical Analysis 1: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Day 1; Test type: Superiority or Other; p = 0.099, Mixed Models Analysis; LS Mean Difference = -5.6, 90% CI 2-sided [-11.1 to 0.0], Standard Error of Mean 2.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Day 10; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis; LS Mean Difference = -5.9, 90% CI 2-sided [-10.1 to -1.7], Standard Error of Mean 2.1 — Difference is MK-8150 dose - placebo

12. Primary Outcome: Change From Baseline in TWA0-24hrs HR in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel H)
Description: HR was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all HR values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each HR value by that HR value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified HR value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value (determined separately in each period).
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel H - MK-8150 10/20 mg | Panel H - Placebo
Number analyzed (Participants) | 7 | 8
beats per minute
  Day 1 (N = 7, 8) | -2.4 (1.3) | 0.0 (2.3)
  Day 10 (N = 6, 8) | -0.6 (1.4) | -2.0 (1.5)
Statistical Analysis 1: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Day 1; Test type: Superiority or Other; p = 0.281, Mixed Models Analysis; LS Mean Difference = -2.4, 90% CI 2-sided [-6.5 to 1.6], Standard Error of Mean 2.0 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Day 10; Test type: Superiority or Other; p = 0.333, Mixed Models Analysis; LS Mean Difference = 1.4, 90% CI 2-sided [-1.2 to 4.0], Standard Error of Mean 1.3 — Difference is MK-8150 dose - placebo

13. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel I)
Description: as for outcome 3
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel I - Placebo: Placebo once daily on Days 1-28
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel I - Placebo
Number analyzed (Participants) | 12 | 6
mm Hg
  Day 1 (N = 12, 6) | -11.2 (1.6) | -7.4 (2.9)
  Day 28 (N = 10, 6) | -15.2 (2.3) | -14.4 (2.6)
Statistical Analysis 1: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 1; Test type: Superiority or Other; p = 0.279, Mixed Models Analysis; LS Mean Difference = -3.8, 90% CI 2-sided [-9.7 to 2.1], Standard Error of Mean 3.4 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 28; Test type: Superiority or Other; p = 0.817, Mixed Models Analysis; LS Mean Difference = -0.8, 90% CI 2-sided [-6.9 to 5.2], Standard Error of Mean 3.4 — Difference is MK-8150 dose - placebo

14. Primary Outcome: Change From Baseline in TWA0-24hrs HR in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel I)
Description: as for outcome 4
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel I - Placebo
Number analyzed (Participants) | 12 | 6
beats per minute
  Day 1 (N = 12, 6) | 0.3 (1.9) | -0.5 (1.4)
  Day 8 (N = 12, 6) | 1.2 (1.9) | -2.8 (2.0)
  Day 15 (N = 10, 6) | 0.8 (2.3) | -1.6 (1.8)
  Day 22 (N = 10, 6) | 0.1 (2.0) | -2.9 (1.4)
  Day 28 (N = 10, 6) | 0.7 (2.7) | -4.4 (1.3)
Statistical Analysis 1: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 1; Test type: Superiority or Other; p = 0.756, Mixed Models Analysis; LS Mean Difference = 0.7, 90% CI 2-sided [-3.2 to 4.7], Standard Error of Mean 2.4 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 8; Test type: Superiority or Other; p = 0.158, Mixed Models Analysis; LS Mean Difference = 3.9, 90% CI 2-sided [-0.7 to 8.6], Standard Error of Mean 2.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 15; Test type: Superiority or Other; p = 0.404, Mixed Models Analysis; LS Mean Difference = 2.4, 90% CI 2-sided [-2.4 to 7.1], Standard Error of Mean 2.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 22; Test type: Superiority or Other; p = 0.214, Mixed Models Analysis; LS Mean Difference = 3.0, 90% CI 2-sided [-1.0 to 7.1], Standard Error of Mean 2.4 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 28; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis; LS Mean Difference = 5.1, 90% CI 2-sided [0.2 to 10.0], Standard Error of Mean 2.9 — Difference is MK-8150 dose - placebo

15. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel J)
Description: as for outcome 3
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel J - Placebo: Placebo once daily on Days 1-28
Arm/Group | Panel J - MK-8150 10/20 mg | Panel J - Placebo
Number analyzed (Participants) | 12 | 6
mm Hg
  Day 1 (N = 12, 6) | -16.7 (2.4) | -5.4 (1.6)
  Day 28 (N = 9, 6) | -11.5 (2.4) | -5.4 (2.4)
Statistical Analysis 1: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 1; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; LS Mean Difference = -11.3, 90% CI 2-sided [-16.8 to -5.9], Standard Error of Mean 3.1 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 28; Test type: Superiority or Other; p = 0.105, Mixed Models Analysis; LS Mean Difference = -6.1, 90% CI 2-sided [-12.3 to 0.1], Standard Error of Mean 3.5 — Difference is MK-8150 dose - placebo

16. Primary Outcome: Change From Baseline in TWA0-24hrs HR in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel J)
Description: as for outcome 4
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel J - MK-8150 10/20 mg | Panel J - Placebo
Number analyzed (Participants) | 12 | 6
beats per minute
  Day 1 (N = 12, 6) | -3.0 (1.1) | -1.6 (3.4)
  Day 8 (N = 11, 6) | -0.6 (1.5) | -2.8 (3.6)
  Day 15 (N = 10, 6) | -1.2 (1.6) | -2.6 (3.0)
  Day 22 (N = 9, 6) | -1.0 (1.5) | 2.0 (4.5)
  Day 28 (N = 9, 6) | -0.3 (1.7) | -2.8 (3.6)
Statistical Analysis 1: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 1; Test type: Superiority or Other; p = 0.691, Mixed Models Analysis; LS Mean Difference = -1.4, 90% CI 2-sided [-7.5 to 4.6], Standard Error of Mean 3.6 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 8; Test type: Superiority or Other; p = 0.570, Mixed Models Analysis; LS Mean Difference = 2.2, 90% CI 2-sided [-4.3 to 8.8], Standard Error of Mean 3.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 15; Test type: Superiority or Other; p = 0.666, Mixed Models Analysis; LS Mean Difference = 1.5, 90% CI 2-sided [-4.2 to 7.1], Standard Error of Mean 3.4 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 22; Test type: Superiority or Other; p = 0.534, Mixed Models Analysis; LS Mean Difference = -3.0, 90% CI 2-sided [-10.9 to 4.9], Standard Error of Mean 4.7 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 28; Test type: Superiority or Other; p = 0.528, Mixed Models Analysis; LS Mean Difference = 2.5, 90% CI 2-sided [-4.1 to 9.2], Standard Error of Mean 4.0 — Difference is MK-8150 dose - placebo

17. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC0-24) of MK-8150 in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel A/B/C/D)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. AUC0-24 of MK-8150 on Day 1 and Day 10 was determined.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
μM*hr
  Day 1 (N = 6, 6, 6, 5) | 1.84 (13) | 3.22 (21) | 6.97 (19) | 5.16 (18)
  Day 10 (N = 5, 6, 4, 5) | 6.76 (36) | 12.3 (30) | 19.2 (23) | 16.1 (34)

18. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of MK-8150 in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel A/B/C/D)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Cmax of MK-8150 on Day 1 and Day 10 was determined from the observed plasma concentration-time data.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose, and (for Day 10 only) 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
μM
  Day 1 (N = 6, 6, 6, 5) | 0.183 (7.7) | 0.353 (18) | 0.656 (12) | 0.502 (32)
  Day 10 (N = 5, 6, 4, 5) | 0.440 (20) | 0.784 (26) | 1.25 (16) | 1.14 (35)

19. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of MK-8150 in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel A/B/C/D)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Tmax of MK-8150 on Day 1 and Day 10 was determined from the observed plasma concentration-time data.
Time Frame: as for outcome 18
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Median (Full Range); unit: hr
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
hr
  Day 1 (N = 6, 6, 6, 5) | 1 (2.6) [0.5 to 1.5] | 1 (2.4) [1 to 2] | 1.25 (2.4) [0.5 to 2] | 1 (2.3) [0.5 to 1.5]
  Day 10 (N = 5, 6, 4, 5) | 1 (3.4) [0.5 to 1.5] | 0.75 (1.0) [0.5 to 2] | 1.25 (1.9) [0.5 to 1.5] | 0.5 (3.7) [0.5 to 1.5]

20. Primary Outcome: Apparent Terminal Half-life (t1/2) of MK-8150 Determined Following Day 10 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel A/B/C/D)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. t1/2 is the time it takes for the concentration of the drug in the body to decrease by half during the elimination phase. t1/2 of MK-8150 was determined from plasma drug concentration data obtained following the last dose of study drug, administered on Day 10.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg
Number analyzed (Participants) | 5 | 6 | 4 | 5
hr | 70.7 (41) | 78.6 (19) | 46.7 (74) | 58.0 (45)

21. Primary Outcome: AUC0-24 of MK-8150 in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 (Panel E/F, Day 1 Dose)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. AUC0-24 of MK-8150 on Day 1 was determined.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Groups:
- Panel E - MK-8150 3 mg Single Dose: Single dose of MK-8150 3 mg administered on Day 1 in Panel E. No drug was administered on Days 2-5
- Panel F - MK-8150 6 mg Single Dose: Single dose of MK-8150 6 mg administered on Day 1 in Panel F. No drug was administered on Days 2-5
Arm/Group | Panel E - MK-8150 3 mg Single Dose | Panel F - MK-8150 6 mg Single Dose
Number analyzed (Participants) | 6 | 6
μM*hr | 1.17 (14) | 2.37 (14)

22. Primary Outcome: Cmax of MK-8150 in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 (Panel E/F, Day 1 Dose)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Cmax of MK-8150 on Day 1 was determined from the observed plasma concentration-time data.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel E - MK-8150 3 mg Single Dose | Panel F - MK-8150 6 mg Single Dose
Number analyzed (Participants) | 6 | 6
μM | 0.129 (25) | 0.268 (17)

23. Primary Outcome: Tmax of MK-8150 in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 (Panel E/F, Day 1 Dose)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Tmax of MK-8150 on Day 1 was determined from the observed plasma concentration-time data.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Median (Full Range); unit: hr
Arm/Group | Panel E - MK-8150 3 mg Single Dose | Panel F - MK-8150 6 mg Single Dose
Number analyzed (Participants) | 6 | 6
hr | 1 (2.6) [1 to 1.5] | 1 (2.4) [0.5 to 1]

24. Primary Outcome: t1/2 of MK-8150 in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 (Panel E/F, Day 1 Dose)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. t1/2 is the time it takes for the concentration of the drug in the body to decrease by half during the elimination phase. t1/2 of MK-8150 was determined from plasma drug concentration data obtained following the Day 1 dose.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel E - MK-8150 3 mg Single Dose | Panel F - MK-8150 6 mg Single Dose
Number analyzed (Participants) | 6 | 6
hr | 85.0 (35) | 82.1 (53)

25. Primary Outcome: AUC0-24 of MK-8150 in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel E/F, Days 6-15)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. AUC0-24 of MK-8150 on Day 6 and Day 15 was determined.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Groups:
- Panel E - MK-8150 2 mg Multiple Dose Administration: Multiple dose administration of MK-8150 2 mg once daily on Days 6-15 in Panel E
- Panel F - MK-8150 4 mg Multiple Dose Administration: Multiple dose administration of MK-8150 4 mg once daily on Days 6-15 in Panel F
Arm/Group | Panel E - MK-8150 2 mg Multiple Dose Administration | Panel F - MK-8150 4 mg Multiple Dose Administration
Number analyzed (Participants) | 5 | 6
μM*hr
  Day 6 (N = 5, 6) | 1.08 (16) | 2.23 (16)
  Day 15 (N = 5, 4) | 2.98 (22) | 6.58 (26)

26. Primary Outcome: Cmax of MK-8150 in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel E/F, Days 6-15)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Cmax of MK-8150 on Day 6 and Day 15 was determined from the observed plasma concentration-time data.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose, and (for Day 15 only) 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel E - MK-8150 2 mg Multiple Dose Administration | Panel F - MK-8150 4 mg Multiple Dose Administration
Number analyzed (Participants) | 5 | 6
μM
  Day 6 (N = 5, 6) | 0.109 (19) | 0.208 (10)
  Day 15 (N = 5, 4) | 0.192 (16) | 0.425 (25)

27. Primary Outcome: Tmax of MK-8150 in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel E/F, Days 6-15)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Tmax of MK-8150 on Day 6 and Day 15 was determined from the observed plasma concentration-time data.
Time Frame: as for outcome 26
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Median (Full Range); unit: hr
Arm/Group | Panel E - MK-8150 2 mg Multiple Dose Administration | Panel F - MK-8150 4 mg Multiple Dose Administration
Number analyzed (Participants) | 5 | 6
hr
  Day 6 (N = 5, 6) | 1 (2.6) [0.5 to 1] | 1 (2.4) [0.5 to 1]
  Day 15 (N = 5, 4) | 1 [0.5 to 1.5] | 1 [1 to 1.5]

28. Primary Outcome: t1/2 of MK-8150 Determined Following Day 15 Dose in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel E/F, Days 6-15)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. t1/2 is the time it takes for the concentration of the drug in the body to decrease by half during the elimination phase. t1/2 of MK-8150 was determined from plasma drug concentration data obtained following the last dose of study drug, administered on Day 15.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel E - MK-8150 2 mg Multiple Dose Administration | Panel F - MK-8150 4 mg Multiple Dose Administration
Number analyzed (Participants) | 5 | 4
hr | 68.1 (36) | 92.6 (63)

29. Primary Outcome: AUC0-24 of MK-8150 in Healthy Male Participants Administered Multiple Doses of MK-8150 (Panel G)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. AUC0-24 of MK-8150 on Day 1 and Day 28 was determined.
Time Frame: Day 1: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose; Day 28: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Arm/Group | Panel G - MK-8150 20/30/40/60 mg
Number analyzed (Participants) | 8
μM*hr
  Day 1 (N = 8) | 8.08 (23)
  Day 28 (N = 7) | 65.5 (30)

30. Primary Outcome: Cmax of MK-8150 in Healthy Male Participants Administered Multiple Doses of MK-8150 (Panel G)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Cmax of MK-8150 on Day 1 and Day 28 was determined from the observed plasma concentration-time data.
Time Frame: Day 1: Pre-dose and 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post dose; Day 28: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel G - MK-8150 20/30/40/60 mg
Number analyzed (Participants) | 8
μM
  Day 1 (N = 8) | 0.664 (8.5)
  Day 28 (N = 7) | 4.05 (22)

31. Primary Outcome: Tmax of MK-8150 in Healthy Male Participants Administered Multiple Doses of MK-8150 (Panel G)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. Tmax of MK-8150 on Day 1 and Day 28 was determined from the observed plasma concentration-time data.
Time Frame: as for outcome 30
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Median (Full Range); unit: hr
Arm/Group | Panel G - MK-8150 20/30/40/60 mg
Number analyzed (Participants) | 8
hr
  Day 1 (N = 8) | 1.0 (2.6) [0.5 to 4]
  Day 28 (N = 7) | 1.5 [1 to 2]

32. Primary Outcome: t1/2 of MK-8150 Determined Following Day 28 Dose in Healthy Male Participants Administered Multiple Doses of MK-8150 (Panel G)
Description: Serial plasma samples for determination of PK parameters were obtained from study participants. t1/2 is the time it takes for the concentration of the drug in the body to decrease by half during the elimination phase. t1/2 of MK-8150 was determined from plasma drug concentration data obtained following the last dose of study drug, administered on Day 28.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel G - MK-8150 20/30/40/60 mg
Number analyzed (Participants) | 7
hr | 51.8 (48)

33. Primary Outcome: AUC0-24 of MK-8150 in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 (Panel H)
Description: as for outcome 17
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Arm/Group | Panel H - MK-8150 10/20 mg
Number analyzed (Participants) | 8
μM*hr
  Day 1 (N = 8) | 3.56 (20)
  Day 10 (N = 6) | 25.1 (31)

34. Primary Outcome: Cmax of MK-8150 in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 (Panel H)
Description: as for outcome 18
Time Frame: as for outcome 18
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel H - MK-8150 10/20 mg
Number analyzed (Participants) | 8
μM
  Day 1 (N = 8) | 0.395 (27)
  Day 10 (N = 6) | 1.71 (31)

35. Primary Outcome: Tmax of MK-8150 in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 (Panel H)
Description: as for outcome 19
Time Frame: as for outcome 18
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Median (Full Range); unit: hr
Arm/Group | Panel H - MK-8150 10/20 mg
Number analyzed (Participants) | 8
hr
  Day 1 (N = 8) | 1.0 (2.6) [0.5 to 2]
  Day 10 (N = 6) | 1.0 [0.5 to 1]

36. Primary Outcome: t1/2 of MK-8150 Determined Following Day 10 Dose in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 (Panel H)
Description: as for outcome 20
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel H - MK-8150 10/20 mg
Number analyzed (Participants) | 6
hr | 69.6 (44)

37. Primary Outcome: AUC0-24 of MK-8150 in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel I/J, Including Only Participants Who Completed Treatment)
Description: as for outcome 29
Time Frame: as for outcome 29
Population: All participants who met protocol entry criteria, received study drug and completed the 28 days of treatment, and had data available for the measure
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel J - MK-8150 10/20 mg
Number analyzed (Participants) | 10 | 9
μM*hr
  Day 1 (N = 10, 9) | 1.80 (19) | 3.80 (16)
  Day 28 (N = 10, 9) | 39.1 (31) | 28.5 (40)

38. Primary Outcome: Cmax of MK-8150 in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel I/J, Including Only Participants Who Completed Treatment)
Description: as for outcome 30
Time Frame: as for outcome 30
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel J - MK-8150 10/20 mg
Number analyzed (Participants) | 10 | 9
μM
  Day 1 (N = 10, 9) | 0.213 (28) | 0.395 (18)
  Day 28 (N = 10, 9) | 2.72 (29) | 1.75 (34)

39. Primary Outcome: Tmax of MK-8150 in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel I/J, Including Only Participants Who Completed Treatment)
Description: as for outcome 31
Time Frame: as for outcome 30
Population: as for outcome 37
Measure: Median (Full Range); unit: hr
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel J - MK-8150 10/20 mg
Number analyzed (Participants) | 10 | 9
hr
  Day 1 (N = 10, 9) | 0.75 (2.6) [0.5 to 2] | 1.0 (2.4) [0.5 to 1]
  Day 28 (N = 10, 9) | 0.5 [0.5 to 1] | 1 [0.5 to 2]

40. Primary Outcome: t1/2 of MK-8150 Determined Following Day 28 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 (Panel I/J, Including Only Participants Who Completed Treatment)
Description: as for outcome 32
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours post dose
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel J - MK-8150 10/20 mg
Number analyzed (Participants) | 10 | 9
hr | 73.9 (37) | 81.0 (18)

41. Secondary Outcome: Change From Baseline in TWA0-24hrs AIx in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel A/B/C/D)
Description: AIx was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Augmentation index is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. Time-weighted average was obtained as follows: For all AIx values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each AIx value by that AIx value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified AIx value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. AIx was adjusted for HR. Baseline was Day 1 pre-dose value.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel A/B/C/D - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8
percentage of central pulse pressure
  Day 1 (N = 6, 6, 6, 5, 8) | -3.7 (1.7) | -9.3 (0.5) | -11.7 (3.3) | -7.2 (1.5) | -3.3 (1.0)
  Day 10 (N = 5, 6, 4, 5, 8) | -2.3 (1.4) | -9.9 (2.1) | -10.9 (1.7) | -5.8 (1.9) | -5.4 (1.4)
Statistical Analysis 1: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.848, Mixed Models Analysis; LS Mean Difference = -0.4, 90% CI 2-sided [-3.8 to 3.0], Standard Error of Mean 2.0 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -6.0, 90% CI 2-sided [-8.0 to -4.0], Standard Error of Mean 1.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; LS Mean Difference = -8.4, 90% CI 2-sided [-14.4 to -2.4], Standard Error of Mean 3.5 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Day 1; Test type: Superiority or Other; p = 0.044, Mixed Models Analysis; LS Mean Difference = -3.9, 90% CI 2-sided [-7.0 to -0.8], Standard Error of Mean 1.8 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.139, Mixed Models Analysis; LS Mean Difference = 3.1, 90% CI 2-sided [-0.4 to 6.6], Standard Error of Mean 2.0 — Difference is MK-8150 dose - placebo
Statistical Analysis 6: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.088, Mixed Models Analysis; LS Mean Difference = -4.5, 90% CI 2-sided [-8.9 to -0.2], Standard Error of Mean 2.5 — Difference is MK-8150 dose - placebo
Statistical Analysis 7: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; LS Mean Difference = -5.5, 90% CI 2-sided [-9.3 to -1.6], Standard Error of Mean 2.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 8: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Day 10; Test type: Superiority or Other; p = 0.878, Mixed Models Analysis; LS Mean Difference = -0.4, 90% CI 2-sided [-4.5 to 3.8], Standard Error of Mean 2.4 — Difference is MK-8150 dose - placebo

42. Secondary Outcome: Change From Baseline in TWA0-24hrs cDBP Following Day 10 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel A/B/C/D)
Description: cDBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cDBP value by that cDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel A/B/C/D - Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 5 | 8
mm Hg | -3.5 (2.4) | -8.1 (1.9) | -9.9 (1.8) | -7.8 (3.0) | -5.7 (2.3)
Statistical Analysis 1: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.512, Mixed Models Analysis; LS Mean Difference = 2.2, 90% CI 2-sided [-3.4 to 7.7], Standard Error of Mean 3.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.429, Mixed Models Analysis; LS Mean Difference = -2.4, 90% CI 2-sided [-7.5 to 2.7], Standard Error of Mean 3.0 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.166, Mixed Models Analysis; LS Mean Difference = -4.2, 90% CI 2-sided [-9.3 to 0.8], Standard Error of Mean 2.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.591, Mixed Models Analysis; LS Mean Difference = -2.1, 90% CI 2-sided [-8.6 to 4.5], Standard Error of Mean 3.8 — Difference is MK-8150 dose - placebo

43. Secondary Outcome: Change From Baseline in TWA0-24hrs pSBP Following Day 10 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel A/B/C/D)
Description: pSBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pSBP value by that pSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel A/B/C/D - Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 5 | 8
mm Hg | -4.5 (3.6) | -10.6 (1.7) | -15.3 (1.2) | -9.0 (2.9) | -10.0 (2.6)
Statistical Analysis 1: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.248, Mixed Models Analysis; LS Mean Difference = 5.5, 90% CI 2-sided [-2.5 to 13.5], Standard Error of Mean 4.7 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.836, Mixed Models Analysis; LS Mean Difference = -0.6, 90% CI 2-sided [-5.6 to 4.4], Standard Error of Mean 2.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.109, Mixed Models Analysis; LS Mean Difference = -5.3, 90% CI 2-sided [-10.7 to 0.1], Standard Error of Mean 3.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.785, Mixed Models Analysis; LS Mean Difference = 1.0, 90% CI 2-sided [-5.4 to 7.5], Standard Error of Mean 3.7 — Difference is MK-8150 dose - placebo

44. Secondary Outcome: Change From Baseline in TWA0-24hrs pDBP Following Day 10 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel A/B/C/D)
Description: pDBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pDBP value by that pDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel A/B/C/D - Placebo
Number analyzed (Participants) | 5 | 6 | 4 | 5 | 8
mm Hg | -2.9 (2.3) | -8.2 (2.1) | -13.6 (2.5) | -8.1 (2.3) | -5.8 (2.1)
Statistical Analysis 1: Comparison: Panel A - MK-8150 5 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.365, Mixed Models Analysis; LS Mean Difference = 2.9, 90% CI 2-sided [-2.5 to 8.3], Standard Error of Mean 3.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 10 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.424, Mixed Models Analysis; LS Mean Difference = -2.4, 90% CI 2-sided [-7.4 to 2.6], Standard Error of Mean 2.9 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 20 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; LS Mean Difference = -7.8, 90% CI 2-sided [-13.3 to -2.2], Standard Error of Mean 3.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 15 mg vs Panel A/B/C/D - Placebo; Test type: Superiority or Other; p = 0.475, Mixed Models Analysis; LS Mean Difference = -2.2, 90% CI 2-sided [-7.5 to 3.0], Standard Error of Mean 3.1 — Difference is MK-8150 dose - placebo

45. Secondary Outcome: Change From Baseline in TWA0-24hrs AIx in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel E)
Description: AIx was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Augmentation index is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. Time-weighted average was obtained as follows: For all AIx values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each AIx value by that AIx value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified AIx value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. AIx was adjusted for HR. Baseline for Day 1 was Day 1 pre-dose value; Baseline for Day 6-15 was Day 6 pre-dose value.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel E - MK-8150 3/2 mg | Panel E - Placebo
Number analyzed (Participants) | 6 | 3
percentage of central pulse pressure
  Day 1 (N = 6, 3) | -3.8 (2.7) | -2.6 (0.9)
  Day 6 (N = 5, 3) | -5.2 (3.6) | -1.0 (0.8)
  Day 15 (N = 5, 3) | -3.5 (2.6) | 0.3 (1.2)
Statistical Analysis 1: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 1; Test type: Superiority or Other; p = 0.715, Mixed Models Analysis; LS Mean Difference = -1.3, 90% CI 2-sided [-7.4 to 4.8], Standard Error of Mean 3.4 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 6; Test type: Superiority or Other; p = 0.338, Mixed Models Analysis; LS Mean Difference = -4.3, 90% CI 2-sided [-11.9 to 3.4], Standard Error of Mean 4.3 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Day 15; Test type: Superiority or Other; p = 0.281, Mixed Models Analysis; LS Mean Difference = -3.9, 90% CI 2-sided [-10.0 to 2.3], Standard Error of Mean 3.4 — Difference is MK-8150 dose - placebo

46. Secondary Outcome: Change From Baseline in TWA0-24hrs cDBP Following Day 15 Dose in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel E)
Description: cDBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cDBP value by that cDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline for Day 1 was Day 1 pre-dose value; Baseline for Day 6-15 was Day 6 pre-dose value.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel E - MK-8150 3/2 mg | Panel E - Placebo
Number analyzed (Participants) | 5 | 3
mm Hg | -5.7 (1.5) | -8.7 (2.4)
Statistical Analysis 1: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Test type: Superiority or Other; p = 0.317, Mixed Models Analysis; LS Mean Difference = 2.9, 90% CI 2-sided [-2.1 to 7.9], Standard Error of Mean 2.8 — Difference is MK-8150 dose - placebo

47. Secondary Outcome: Change From Baseline in TWA0-24hrs pSBP Following Day 15 Dose in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel E)
Description: pSBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pSBP value by that pSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline for Day 1 was Day 1 pre-dose value; Baseline for Day 6-15 was Day 6 pre-dose value.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel E - MK-8150 3/2 mg | Panel E - Placebo
Number analyzed (Participants) | 5 | 3
mm Hg | -0.4 (3.5) | -7.1 (1.3)
Statistical Analysis 1: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Test type: Superiority or Other; p = 0.090, Mixed Models Analysis; LS Mean Difference = 6.7, 90% CI 2-sided [0.2 to 13.2], Standard Error of Mean 3.6 — Difference is MK-8150 dose - placebo

48. Secondary Outcome: Change From Baseline in TWA0-24hrs pDBP Following Day 15 Dose in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel E)
Description: pDBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pDBP value by that pDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline for Day 1 was Day 1 pre-dose value; Baseline for Day 6-15 was Day 6 pre-dose value.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel E - MK-8150 3/2 mg | Panel E - Placebo
Number analyzed (Participants) | 5 | 3
mm Hg | -0.9 (1.5) | -4.1 (1.4)
Statistical Analysis 1: Comparison: Panel E - MK-8150 3/2 mg vs Panel E - Placebo; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis; LS Mean Difference = 3.3, 90% CI 2-sided [-0.3 to 6.8], Standard Error of Mean 2.0 — Difference is MK-8150 dose - placebo

49. Secondary Outcome: Change From Baseline in TWA0-24hrs AIx in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel F)
Description: as for outcome 45
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel F - MK-8150 6/4 mg | Panel F - Placebo
Number analyzed (Participants) | 6 | 3
percentage of central pulse pressure
  Day 1 (N = 6, 3) | -4.8 (2.3) | -2.5 (2.1)
  Day 6 (N = 6, 3) | -5.1 (1.5) | 0.5 (2.6)
  Day 15 (N = 4, 3) | -6.8 (2.1) | 0.9 (2.2)
Statistical Analysis 1: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 1; Test type: Superiority or Other; p = 0.477, Mixed Models Analysis; LS Mean Difference = -2.3, 90% CI 2-sided [-7.9 to 3.3], Standard Error of Mean 3.1 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 6; Test type: Superiority or Other; p = 0.090, Mixed Models Analysis; LS Mean Difference = -5.6, 90% CI 2-sided [-11.0 to -0.2], Standard Error of Mean 3.0 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Day 15; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis; LS Mean Difference = -7.6, 90% CI 2-sided [-13.0 to -2.2], Standard Error of Mean 3.0 — Difference is MK-8150 dose - placebo

50. Secondary Outcome: Change From Baseline in TWA0-24hrs cDBP Following Day 15 Dose in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel F)
Description: as for outcome 46
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel F - MK-8150 6/4 mg | Panel F - Placebo
Number analyzed (Participants) | 4 | 3
mm Hg | -10.0 (2.0) | -9.6 (1.6)
Statistical Analysis 1: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Test type: Superiority or Other; p = 0.877, Mixed Models Analysis; LS Mean Difference = -0.4, 90% CI 2-sided [-4.9 to 4.1], Standard Error of Mean 2.5 — Difference is MK-8150 dose - placebo

51. Secondary Outcome: Change From Baseline in TWA0-24hrs pSBP Following Day 15 Dose in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel F)
Description: as for outcome 47
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel F - MK-8150 6/4 mg | Panel F - Placebo
Number analyzed (Participants) | 4 | 3
mm Hg | -12.8 (2.8) | -11.7 (3.2)
Statistical Analysis 1: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Test type: Superiority or Other; p = 0.827, Mixed Models Analysis; LS Mean Difference = -1.0, 90% CI 2-sided [-9.3 to 7.2], Standard Error of Mean 4.6 — Difference is MK-8150 dose - placebo

52. Secondary Outcome: Change From Baseline in TWA0-24hrs pDBP Following Day 15 Dose in Elderly Male and Female Participants With Mild to Moderate Hypertension Administered Single and Multiple Doses of MK-8150 and Placebo (Panel F)
Description: as for outcome 48
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel F - MK-8150 6/4 mg | Panel F - Placebo
Number analyzed (Participants) | 4 | 3
mm Hg | -9.3 (1.7) | -4.1 (2.9)
Statistical Analysis 1: Comparison: Panel F - MK-8150 6/4 mg vs Panel F - Placebo; Test type: Superiority or Other; p = 0.161, Mixed Models Analysis; LS Mean Difference = -5.2, 90% CI 2-sided [-11.4 to 1.0], Standard Error of Mean 3.5 — Difference is MK-8150 dose - placebo

53. Secondary Outcome: Change From Baseline in TWA0-24hrs AIx in Healthy Male Participants Administered Multiple Doses of MK-8150 and Placebo (Panel G)
Description: as for outcome 41
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel G - MK-8150 20/30/40/60 mg | Panel G - Placebo
Number analyzed (Participants) | 8 | 2
percentage of central pulse pressure
  Day 1 (N = 8, 2) | -11.8 (2.1) | -1.3 (3.8)
  Day 28 (N = 7, 2) | -14.2 (2.1) | -1.4 (0.5)
Statistical Analysis 1: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 1; Test type: Superiority or Other; p = 0.046, Mixed Models Analysis; LS Mean Difference = -10.5, 90% CI 2-sided [-18.8 to -2.3], Standard Error of Mean 4.4 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Day 28; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference = -12.9, 90% CI 2-sided [-17.2 to -8.6], Standard Error of Mean 2.3 — Difference is MK-8150 dose - placebo

54. Secondary Outcome: Change From Baseline in TWA0-24hrs cDBP Following Day 28 Dose in Healthy Male Participants Administered Multiple Doses of MK-8150 and Placebo (Panel G)
Description: as for outcome 42
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel G - MK-8150 20/30/40/60 mg | Panel G - Placebo
Number analyzed (Participants) | 7 | 2
mm Hg | -5.3 (1.7) | -5.6 (1.4)
Statistical Analysis 1: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Test type: Superiority or Other; p = 0.910, Mixed Models Analysis; LS Mean Difference = 0.3, 90% CI 2-sided [-4.6 to 5.2], Standard Error of Mean 2.6 — Difference is MK-8150 dose - placebo

55. Secondary Outcome: Change From Baseline in TWA0-24hrs pSBP Following Day 28 Dose in Healthy Male Participants Administered Multiple Doses of MK-8150 and Placebo (Panel G)
Description: as for outcome 43
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel G - MK-8150 20/30/40/60 mg | Panel G - Placebo
Number analyzed (Participants) | 7 | 2
mm Hg | -6.9 (2.5) | -6.5 (2.1)
Statistical Analysis 1: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Test type: Superiority or Other; p = 0.906, Mixed Models Analysis; LS Mean Difference = -0.4, 90% CI 2-sided [-6.6 to 5.7], Standard Error of Mean 3.6 — Difference is MK-8150 dose - placebo

56. Secondary Outcome: Change From Baseline in TWA0-24hrs pDBP Following Day 28 Dose in Healthy Male Participants Administered Multiple Doses of MK-8150 and Placebo (Panel G)
Description: as for outcome 44
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel G - MK-8150 20/30/40/60 mg | Panel G - Placebo
Number analyzed (Participants) | 7 | 2
mm Hg | -6.5 (1.6) | -6.1 (1.1)
Statistical Analysis 1: Comparison: Panel G - MK-8150 20/30/40/60 mg vs Panel G - Placebo; Test type: Superiority or Other; p = 0.870, Mixed Models Analysis; LS Mean Difference = -0.4, 90% CI 2-sided [-4.4 to 3.7], Standard Error of Mean 2.4 — Difference is MK-8150 dose - placebo

57. Secondary Outcome: Change From Baseline in TWA0-24hrs AIx in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel H)
Description: AIx was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Augmentation index is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. Time-weighted average was obtained as follows: For all AIx values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each AIx value by that AIx value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified AIx value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. AIx was adjusted for HR. Baseline was Day 1 pre-dose value (determined separately in each period).
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel H - MK-8150 10/20 mg | Panel H - Placebo
Number analyzed (Participants) | 7 | 8
percentage of central pulse pressure
  Day 1 (N = 7, 8) | -3.9 (0.9) | 0.4 (0.9)
  Day 10 (N = 6, 8) | -5.8 (1.3) | 2.4 (1.1)
Statistical Analysis 1: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Day 1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -4.3, 90% CI 2-sided [-5.0 to -3.7], Standard Error of Mean 0.3 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Day 10; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference = -8.2, 90% CI 2-sided [-10.7 to -5.7], Standard Error of Mean 1.2 — Difference is MK-8150 dose - placebo

58. Secondary Outcome: Change From Baseline in TWA0-24hrs cDBP Following Day 10 Dose in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel H)
Description: cDBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cDBP value by that cDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value (determined separately in each period).
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel H - MK-8150 10/20 mg | Panel H - Placebo
Number analyzed (Participants) | 6 | 8
mm Hg | -4.6 (1.8) | -1.8 (1.3)
Statistical Analysis 1: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis; LS Mean Difference = -2.8, 90% CI 2-sided [-4.9 to -0.8], Standard Error of Mean 1.0 — Difference is MK-8150 dose - placebo

59. Secondary Outcome: Change From Baseline in TWA0-24hrs pSBP Following Day 10 Dose in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel H)
Description: pSBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pSBP value by that pSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value (determined separately in each period).
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel H - MK-8150 10/20 mg | Panel H - Placebo
Number analyzed (Participants) | 6 | 8
mm Hg | -15.0 (3.5) | -12.6 (1.8)
Statistical Analysis 1: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Test type: Superiority or Other; p = 0.238, Mixed Models Analysis; LS Mean Difference = -2.4, 90% CI 2-sided [-6.0 to 1.2], Standard Error of Mean 1.8 — Difference is MK-8150 dose - placebo

60. Secondary Outcome: Change From Baseline in TWA0-24hrs pDBP Following Day 10 Dose in Male and Female Participants With Resistant Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel H)
Description: pDBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pDBP value by that pDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. Baseline was Day 1 pre-dose value (determined separately in each period).
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel H - MK-8150 10/20 mg | Panel H - Placebo
Number analyzed (Participants) | 6 | 8
mm Hg | -8.9 (1.8) | -6.3 (1.5)
Statistical Analysis 1: Comparison: Panel H - MK-8150 10/20 mg vs Panel H - Placebo; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis; LS Mean Difference = -2.6, 90% CI 2-sided [-4.7 to -0.6], Standard Error of Mean 1.0 — Difference is MK-8150 dose - placebo

61. Secondary Outcome: Change From Baseline in TWA0-24hrs AIx in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel I)
Description: as for outcome 41
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: percentage of pulse pressure
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel I - Placebo
Number analyzed (Participants) | 12 | 6
percentage of pulse pressure
  Day 1 (N = 12, 6) | -4.9 (1.0) | -4.5 (1.2)
  Day 28 (N = 10, 6) | -10.6 (1.9) | -4.8 (2.1)
Statistical Analysis 1: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 1; Test type: Superiority or Other; p = 0.830, Mixed Models Analysis; LS Mean Difference = -0.4, 90% CI 2-sided [-3.2 to 2.5], Standard Error of Mean 1.6 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Day 28; Test type: Superiority or Other; p = 0.063, Mixed Models Analysis; LS Mean Difference = -5.8, 90% CI 2-sided [-10.8 to -0.7], Standard Error of Mean 2.9 — Difference is MK-8150 dose - placebo

62. Secondary Outcome: Change From Baseline in TWA0-24hrs cDBP Following Day 28 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel I)
Description: as for outcome 42
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel I - Placebo
Number analyzed (Participants) | 10 | 6
mm Hg | -7.7 (1.4) | -7.2 (3.4)
Statistical Analysis 1: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Test type: Superiority or Other; p = 0.892, Mixed Models Analysis; LS Mean Difference = -0.5, 90% CI 2-sided [-7.1 to 6.1], Standard Error of Mean 3.7 — Difference is MK-8150 dose - placebo

63. Secondary Outcome: Change From Baseline in TWA0-24hrs pSBP Following Day 28 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel I)
Description: as for outcome 43
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel I - Placebo
Number analyzed (Participants) | 10 | 6
mm Hg | -12.4 (2.4) | -14.2 (1.8)
Statistical Analysis 1: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis; LS Mean Difference = 1.7, 90% CI 2-sided [-3.4 to 6.9], Standard Error of Mean 3.1 — Difference is MK-8150 dose - placebo

64. Secondary Outcome: Change From Baseline in TWA0-24hrs pDBP Following Day 28 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel I)
Description: as for outcome 44
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel I - MK-8150 5/10/20/40 mg | Panel I - Placebo
Number analyzed (Participants) | 10 | 6
mm Hg | -10.3 (1.4) | -9.6 (2.4)
Statistical Analysis 1: Comparison: Panel I - MK-8150 5/10/20/40 mg vs Panel I - Placebo; Test type: Superiority or Other; p = 0.816, Mixed Models Analysis; LS Mean Difference = -0.7, 90% CI 2-sided [-5.4 to 4.0], Standard Error of Mean 2.8 — Difference is MK-8150 dose - placebo

65. Secondary Outcome: Change From Baseline in TWA0-24hrs AIx Following Day 28 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel J)
Description: as for outcome 41
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel J - MK-8150 10/20 mg | Panel J - Placebo
Number analyzed (Participants) | 12 | 6
percentage of central pulse pressure
  Day 1 (N = 12, 6) | -10.4 (1.8) | -5.9 (1.0)
  Day 28 (N = 9, 6) | -9.9 (2.1) | -6.1 (1.0)
Statistical Analysis 1: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 1; Test type: Superiority or Other; p = 0.061, Mixed Models Analysis; LS Mean Difference = -4.5, 90% CI 2-sided [-8.4 to -0.6], Standard Error of Mean 2.2 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Day 28; Test type: Superiority or Other; p = 0.161, Mixed Models Analysis; LS Mean Difference = -3.8, 90% CI 2-sided [-8.3 to 0.7], Standard Error of Mean 2.6 — Difference is MK-8150 dose - placebo

66. Secondary Outcome: Change From Baseline in TWA0-24hrs cDBP Following Day 28 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel J)
Description: as for outcome 42
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Panel J - MK-8150 10/20 mg | Panel J - Placebo
Number analyzed (Participants) | 9 | 6
mmHg | -4.9 (1.4) | -4.3 (1.5)
Statistical Analysis 1: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Test type: Superiority or Other; p = 0.786, Mixed Models Analysis; LS Mean Difference = -0.5, 90% CI 2-sided [-4.0 to 2.9], Standard Error of Mean 2.0 — Difference is MK-8150 dose - placebo

67. Secondary Outcome: Change From Baseline in TWA0-24hrs pSBP Following Day 28 Dose in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel J)
Description: as for outcome 43
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel J - MK-8150 10/20 mg | Panel J - Placebo
Number analyzed (Participants) | 9 | 6
mm Hg | -9.2 (2.2) | -5.5 (2.2)
Statistical Analysis 1: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Test type: Superiority or Other; p = 0.263, Mixed Models Analysis; LS Mean Difference = -3.8, 90% CI 2-sided [-9.3 to 1.8], Standard Error of Mean 3.3 — Difference is MK-8150 dose - placebo

68. Secondary Outcome: Change From Baseline in TWA0-24hrs pDBP in Male Participants With Mild to Moderate Hypertension Administered Multiple Doses of MK-8150 and Placebo (Panel J)
Description: as for outcome 44
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: All participants who met protocol entry criteria, received study drug and had data available for the measure
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel J - MK-8150 10/20 mg | Panel J - Placebo
Number analyzed (Participants) | 9 | 6
mm Hg | -6.5 (1.3) | -5.3 (1.5)
Statistical Analysis 1: Comparison: Panel J - MK-8150 10/20 mg vs Panel J - Placebo; Test type: Superiority or Other; p = 0.565, Mixed Models Analysis; LS Mean Difference = -1.1, 90% CI 2-sided [-4.4 to 2.1], Standard Error of Mean 2.0 — Difference is MK-8150 dose - placebo

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose (Up to approximately 42 days, excluding pre-dose/screening period)
Description: The 8 crossover Panel H participants are represented in both Panel H - MK-8150 10/20 mg column and Placebo (Panel A - J) column.
Groups:
- Panel J - MK-8150 10/20 mgEdit: MK-8150 once daily as follows: 10 mg (Days 1-7), 20 mg (Days 8-28)
Arm/Group | Panel A - MK-8150 5 mg | Panel B - MK-8150 10 mg | Panel C - MK-8150 20 mg | Panel D - MK-8150 15 mg | Panel E - MK-8150 3/2 mg | Panel F - MK-8150 6/4 mg | Panel G - MK-8150 20/30/40/60 mg | Panel H - MK-8150 10/20 mg | Panel I - MK-8150 5/10/20/40 mg | Panel J - MK-8150 10/20 mgEdit | Placebo (Panel A - J) | Post Study | Screening
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/8 | 0/8 | 0/12 | 0/12 | 0/36 | 0/103 | 0/103
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 6/6 | 3/5 | 4/6 | 3/6 | 7/8 | 6/8 | 12/12 | 10/12 | 23/36 | 1/103 | 11/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A - MK-8150 5 mg (N=6) | Panel B - MK-8150 10 mg (N=6) | Panel C - MK-8150 20 mg (N=6) | Panel D - MK-8150 15 mg (N=5) | Panel E - MK-8150 3/2 mg (N=6) | Panel F - MK-8150 6/4 mg (N=6) | Panel G - MK-8150 20/30/40/60 mg (N=8) | Panel H - MK-8150 10/20 mg (N=8) | Panel I - MK-8150 5/10/20/40 mg (N=12) | Panel J - MK-8150 10/20 mgEdit (N=12) | Placebo (Panel A - J) (N=36) | Post Study (N=103) | Screening (N=103)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Pyrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Common cold (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 6 (6)
Abdominal wall strained (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fasting hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (8) | 1 (1) | 0 (0) | 0 (0)
Pain in leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Dizziness upon standing (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 1 (3) | 2 (3) | 2 (5) | 0 (0) | 4 (15) | 5 (15) | 12 (25) | 4 (36) | 17 (38) | 0 (0) | 1 (1)
Intermittent headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ischialgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Short-term memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis irritant contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczematous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.